CLINICAL TRIAL: NCT01423019
Title: A Comparative Effectiveness Study Evaluating the Effects of Two Thermogenic Supplements on Body Composition Using a Double-Blinded Placebo-Controlled Protocol
Brief Title: A Comparative Effectiveness Study Evaluating the Effects of Thermogenic Supplements on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Health Technologies, Inc. (Network)
Responsible Party: Principal Investigator, Gilbert R Kaats, Dr. Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Nutratech - 60
Record Dates: First submitted 2011-07-05; First posted 2011-08-25 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Weight Loss
Keywords: Weight Loss; Body Composition; Fat Free Mass; Bone Mineral Density; Adipose Tissue; Dual-Energy X-Ray Absorptiometry; Body Fat; Eating and appetite control; Basal Metabolic Rate
MeSH Terms: conditions — Weight Loss | interventions — naringin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Advantra Z (Active Comparator): Proprietary ingredient for: stimulating thermogenesis, reducing weight, increasing lean muscle mass to total body mass, improving athletic performance, and suppressing appetite
  Interventions: Dietary Supplement: Advantra Z
- Advantra Z + Naringin + Hesperiden (Active Comparator)
  Interventions: Dietary Supplement: Advantra Z + Naringin + Hesperiden
- Sugar pill (Placebo Comparator): Capsule contains inert ingredient.
  Interventions: Other: Sugar pill

INTERVENTIONS:
Dietary Supplement: Advantra Z — Two capsules are taken twice daily, 20-30 minutes before breakfast and evening meals. Two capsules contain a total of 50 mg p-synephrine.
  Other Names: p-synephrine
  Arms: Advantra Z
Dietary Supplement: Advantra Z + Naringin + Hesperiden — Two capsules are taken twice daily, 20-30 minutes before breakfast and evening meals. Two capsules contain a total of 50 mg p-synephrine, 600 mg naringin, and 100 mg hesperiden.
  Other Names: Naringin; Hesperiden
  Arms: Advantra Z + Naringin + Hesperiden
Other: Sugar pill — Two capsules containing inert ingredients are taken twice daily, 20-30 minutes before breakfast and evening meals.
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether subjects taking a supplement designed to increase metabolic rate will have a positive effect on body composition (fat mass, muscle mass, and bone density.)

DETAILED DESCRIPTION:
In a previous randomized double-blinded placebo-controlled pilot study, subjects taking the nutritional supplements contained in these two weight loss plans had a short-term statistically significant increase in their resting metabolic rates as compared to taking a placebo. No increases were found in blood pressure, resting heart rate, or self-reported discomfort when taking the supplement.

The current study was designed to extend the findings of the pilot study over a 60-day study period using a randomized double-blinded placebo-controlled protocol with the same weight loss interventions.

ELIGIBILITY:
Inclusion Criteria:

* Must ensure with medical provider that there are no medical conditions that would preclude participation
* Must be able to swallow capsules
* Must be age 21 or above

Exclusion Criteria:

* Pregnant or breast feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Body Composition (fat, fat-free mass and bone mineral density) as measured by Dual Energy X-ray Absorptiometry (DXA) | 0 and 60 days
  This study goes beyond assessing changes in scale weight and BMI. DXA is used to assess changes in body composition (lean, fat and bone) associated with the weight loss interventions.

SECONDARY OUTCOMES:
43-item blood chemistry panel | 0 and 60 days
  43 chemistries including Lipids, CBC, Metabolic panel, TSH, and Cardio CrP
Change from Baseline in Systolic and Diastolic Blood Pressure at 30 days | 0 and 30 days
  Measures the amount of force (pressure) that blood exerts on the walls of the blood vessels as it passes through them. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic pressure is a measure of blood pressure while the heart is relaxed, between heartbeats. Measurements will be taken after sitting or lying down for at least 5 minutes. Changes will be reported between baseline and day 30 of study.
Change from Baseline in Resting Heart Rate at 30 days | 0 and 30 days
  Measure of heart rate after sitting or lying down for at least 5 minutes. Changes will be reported between baseline and day 30 of study.
Change from midpoint of study in Resting Heart Rate at 60 days | 30 and 60 days
  Measure of heart rate after sitting or lying down for at least 5 minutes. Changes will be reported between day 30 and 60 of study.
Change from Baseline in Systolic and Diastolic Blood Pressure at 60 days | 0 and 60 days
  Measures the amount of force (pressure) that blood exerts on the walls of the blood vessels as it passes through them. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic pressure is a measure of blood pressure while the heart is relaxed, between heartbeats. Measurements will be taken after sitting or lying down for at least 5 minutes. Changes will be reported between baseline and day 60 of study.
Change from Baseline in Resting Heart Rate at 60 days | 0 and 60 days
  Measure of heart rate after sitting or lying down for at least 5 minutes. Changes will be reported between baseline and day 60 of study.
Change from Baseline in self-reported quality of life at 30 days. | 0 and 30 days
Change from mid-point of study in self-reported quality of life at 60 days. | 30 and 60 days
Change from Baseline in self-reported quality of life at 60 days. | 0 and 60 days
Change from Baseline in self-reported eating behavior at 30 days. | 0 and 30 days
  A subscale of the 86-item quality of life inventory assessing 15 items related to the subjects' ability to control eating behavior
Change from mid-point of study in self-reported eating behavior at 60 days | 30 and 60 days
  A subscale of the 86-item quality of life inventory assessing 15 items related to the subjects' ability to control eating behavior
Change from Baseline in self-reported eating behavior at 60 days. | 0 and 60 days
  A subscale of the 86-item quality of life inventory assessing 15 items related to the subjects' ability to control eating behavior
Change from mid-point of study in Systolic and Diastolic Blood Pressure at 60 days | 30 and 60 days
  Measures the amount of force (pressure) that blood exerts on the walls of the blood vessels as it passes through them. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic pressure is a measure of blood pressure while the heart is relaxed, between heartbeats. Measurements will be taken after sitting or lying down for at least 5 minutes. Changes will be reported between mid-point and day 60 of study.
Number of participants with adverse events | up to 60 days
  Participants will have opportunity to report on a daily basis any adverse events experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD FACN, Principal Investigator — Integrative Health Technologies, Inc.; Harry G Preuss, MD MACN, Study Chair — Georgetown University Medical Center, Departments of Biochemistry, Medicine and Pathology; Sidney J Stohs, PhD, Study Director — Dean Emeritus, Creighton University Health Sciences Center
Locations (1):
- Integrative Health Technologies, Inc., San Antonio, Texas, United States

REFERENCES:
- [Background] Stohs SJ, Preuss HG, Keith SC, Keith PL, Miller H, Kaats GR. Effects of p-synephrine alone and in combination with selected bioflavonoids on resting metabolism, blood pressure, heart rate and self-reported mood changes. Int J Med Sci. 2011 Apr 28;8(4):295-301. doi: 10.7150/ijms.8.295. PMID 21537493